CLINICAL TRIAL: NCT05329454
Title: An Open-label, Randomized, 3-way Crossover Study to Evaluate the Pharmacokinetics of Investigational Product Ibuprofen Modified-Release Tablets 800 mg Compared to Ibuprofen Tablets 800 mg in Healthy Volunteers
Brief Title: To Evaluate the Food Effect and the Absorption Profile of Ibuprofen Modified-Release Tablets 800 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Overseas Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OVEIBUA20181121
Record Dates: First submitted 2021-02-04; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-12

CONDITIONS: Chronic Pain
Keywords: Ibuprofen Modified-Release Tablets; Overseas Pharmaceuticals; pain relief
MeSH Terms: conditions — Chronic Pain | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: An open label, randomized, single and multiple-dose, test-versus-reference drug, fed-versus-fasted, 3-way crossover study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment ABC (Experimental): Receive the investigational product and active comparator in a sequence of treatment A, treatment B and treatment C.
  Interventions: Drug: Ibuprofen Tablets
- Treatment ACB (Experimental): Receive the investigational product and active comparator in a sequence of treatment A, treatment C and treatment B.
  Interventions: Drug: Ibuprofen Tablets
- Treatment BAC (Experimental): Receive the investigational product and active comparator in a sequence of treatment B, treatment A and treatment C.
  Interventions: Drug: Ibuprofen Tablets
- Treatment BCA (Experimental): Receive the investigational product and active comparator in a sequence of treatment B, treatment C and treatment A.
  Interventions: Drug: Ibuprofen Tablets
- Treatment CAB (Experimental): Receive the investigational product and active comparator in a sequence of treatment C, treatment A and treatment B.
  Interventions: Drug: Ibuprofen Tablets
- Treatment CBA (Experimental): Receive the investigational product and active comparator in a sequence of treatment C, treatment B and treatment A.
  Interventions: Drug: Ibuprofen Tablets

INTERVENTIONS:
Drug: Ibuprofen Tablets — Treatment A:
  One tablet of IBUMR will be administered to the subjects under fasted condition, followed by a minimum of 72-hour washout interval. After the washout period, subjects will receive 1 × IBUMR every 12 hours for a total of 7 doses.
  Treatment B:
  One tablet of IBURed will be administered to the subjects under fasted condition, followed by a minimum of 72-hour washout interval. After the washout period, subjects will receive 1 × IBURed every 8 hours for a total of 10 doses.
  Treatment C:
  Single dose of IBUMR will be given to the subjects under fed condition (a standard high-fat, high calorie breakfast should be consumed within 30 minutes prior to dosing).

SUMMARY:
An open-label, randomized, 3-way crossover study to evaluate the pharmacokinetics of investigational product "Ibuprofen Modified-Release Tablets 800 mg" in comparison to the reference standard "Ibuprofen Regular-Release Tablets 600 mg/800 mg" in normal healthy volunteers

Primary objective:

To evaluate the food effect of IBUMR and its bioavailability of single and multiple doses compared with reference drugs in normal healthy volunteers.

Secondary objectives:

1. To determine and compare the single and multiple dose PK profiles of IBUMR and reference drugs.
2. To identify the effect duration for IBUMR after dose administration by detecting ibuprofen concentrations in plasma.
3. To evaluate the safety profile of single and multiple doses of IBUMR.

DETAILED DESCRIPTION:
This study consists of 3 treatment periods as below. For Treatment A and Treatment B, single- and multiple-dose stages are included.

Treatment A:

One tablet of IBUMR will be administered to the subjects under fasted condition, followed by a minimum of 72-hour washout interval. After the washout period, subjects will receive 1 × IBUMR every 12 hours for a total of 8 doses.

Treatment B:

One tablet of IBURed-800mg will be administered to the subjects under fasted condition, followed by a minimum of 72-hour washout interval. After the washout period, subjects will receive 1 × IBURed-600mg every 8 hours for a total of 12 doses.

Treatment C:

Single dose of IBUMR will be given to the subjects under fed condition (a standard high-fat, high calorie breakfast should be consumed within 30 minutes prior to dosing).

A minimum of 3-day washout interval will be introduced across the 3 treatment periods. Subjects will be required to be fasted for at least 10 hours prior to the administration of morning doses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose body mass index (BMI) at screening is within a range of ≥18.5 kg/m2 and <25.0 kg/m2.

BMI = Body Weight (kg) / [Height (m)]2 And body weight is not less than 50 kg and 45 kg for males and females, respectively.

* Subject's medical history shows no contraindication to the test medications (hypersensitivity to ibuprofen or any component of test and reference products) and non-steroidal anti-inflammatory drugs (NSAIDs).
* Subjects who are judged to be in good health by the investigator based upon the results of physical examination (PE), vital signs, and routine laboratory tests.
* The female subject shows negative pregnancy test results within 30 days prior to the first dose of the study.
* The subject did not take any of the following medications in the specified durations:
* Any systemically absorbed medication within 14 days (excluding vitamins, food supplements and hormone contraceptives not ibuprofen drug interactions) prior to the first dose of the study
* Any enzyme inducer/inhibitor and/or known hepatic or renal clearance-altering agents (e.g., erythromycin, cimetidine, barbiturates, phenothiazine, clarithromycin, troleandomycin, ketoconazole, miconazolem fluconazole, itraconazole) within 30 days prior to the first dose of the study.
* Subjects are willing to comply with protocol-stated requirements, instructions and restrictions, followed by understanding and signing the written informed consent form by the subject or legal representative if he/she is under the statutory age of consent as per the local authority.

Exclusion Criteria:

* Subjects with any properly diagnosed disease within 30 days prior to the first dose of the study.
* Subjects with a clinically significant hematological, endocrine, cardiovascular, hepatic, renal, gastrointestinal, and/or pulmonary disorder; subjects with any predisposing condition that might interfere with the absorption, distribution, metabolism and excretion of drugs; subjects who has had any previous gastrointestinal surgery or coronary artery bypass graft.
* Subjects who require treatment with any medications, either prescription or non-prescription (excluding vitamins and food supplements), within 30 days prior to the first dose of the study
* Subjects have participated in investigational drug trials and took any investigational drug within 60 days prior to the first does of the study.
* Subjects had blood donation more than 250 and 500 mL within 60 and 90 days, respectively prior to the first dose of the study.
* Subjects had a history of drug abuse or alcohol abuse according to the Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV) criteria.
* Subjects cannot stop smoking and caffeine-intakes for 48 hours prior to the first dose of the study and during the entire study period.
* Subjects who are pregnant or lactating.
* Subjects who have been tested positive for the following tests:
* Human immunodeficiency virus (HIV)
* Hepatitis B virus (HBV)
* Hepatitis C virus (HCV)
* Treponema pallidum (STS test)
* For enrollment of female subjects with child-bearing potential, the subject must be practicing sexual abstinence or be using and willing to continue to use a medically acceptable form of birth control for at least 30 days prior to screening (that period will extend to 3 months for oral contraceptive use) and for at least 30 days after the last dose of study drug. For a subject to be considered not to be of child-bearing potential, she must have been amenorrheic for at least 2 years, or must have had a hysterectomy, a bilateral tubal ligation, and/or a bilateral oophorectomy (as determined by the medical history). The male partner of a female study subject with childbearing potential must use a condom and ensure that his partner uses a suitable method of contraception as outlined above.
* Subjects with underlying medical, mental, psychological, or other inappropriate conditions that would impair treatment compliance, or in the opinion of the investigator would not permit to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-07-18 (Actual)

PRIMARY OUTCOMES:
Comparison of single-dose and multiple-dose bioavailability between IBUMR and IBURed | After collecting blood samples from the last participant, up to 30 days
  Comparison of single-dose and multiple-dose bioavailability between IBUMR and IBURed in log-transformed values of area under the curve from time 0 to the last measurable concentration (AUCL)
Comparison of single-dose and multi-dose bioavailability of IBUMR and IBURed | After collecting blood samples from the last participant, up to 30 days
  Comparison of single-dose and multiple-dose bioavailability between IBUMR and IBURed in log-transformed values of the peak concentration (Cmax)
Comparison of single - and multi-dose bioavailability of IBUMR and IBURed | After collecting blood samples from the last participant, up to 30 days
  Comparison of single-dose and multiple-dose bioavailability between IBUMR and IBURed in log-transformed values of area under the curve from time 0 to infinity (AUCinf).
To assess the food effect of IBUMR in the PK parameters | After collecting blood samples from the last participant, up to 30 days
  To assess the food effect of IBUMR in the PK parameters including Cmax
To evaluate the food effect of IBUMR on PK parameters | After collecting blood samples from the last participant, up to 30 days
  To assess the food effect of IBUMR in the PK parameters including time to reach peak concentration (Tmax)
To evaluate the food effects of IBUMR on PK parameters | After collecting blood samples from the last participant, up to 30 days
  To assess the food effect of IBUMR in the PK parameters including AUCL
Evaluate the food effect of IBUMR in PK parameters | After collecting blood samples from the last participant, up to 30 days
  To assess the food effect of IBUMR in the PK parameters including AUCinf
Determine the food effect of IBUMR in PK parameters | After collecting blood samples from the last participant, up to 30 days
  To assess the food effect of IBUMR in the PK parameters including elimination half-life (t1/2)

SECONDARY OUTCOMES:
Single-dose PK measures | After collecting blood samples from the last participant, up to 30 days
  -- Time to reach peak concentration (Tmax)
Single dose PK method | After collecting blood samples from the last participant, up to 30 days
  -- Area under the concentration-time curve within time span t1 to t2 (AUCt1→t2)
Single dose PK | After collecting blood samples from the last participant, up to 30 days
  -- Area under the concentration-time curve extrapolated from the last detectable sampling time point to infinity as a percentage of total AUC (AUCextrap)
Single dose PK step | After collecting blood samples from the last participant, up to 30 days
  -- Elimination half-life (t1/2)
Single dose PK design | After collecting blood samples from the last participant, up to 30 days
  -- Apparent oral clearance (CL/F)
Single dose PK moves | After collecting blood samples from the last participant, up to 30 days
  -- Apparent volume of distribution after oral administration (Vd/F)
Multiple-dose PK measures | After collecting blood samples from the last participant, up to 30 days
  -- Peak concentration at steady state (Cmax,ss)
Multiple - dosed PK | After collecting blood samples from the last participant, up to 30 days
  -- Plasma drug concentration at a specified time t steady state (Ct,ss)
Multiple - dosed PK method | After collecting blood samples from the last participant, up to 30 days
  -- Average concentration at steady state (Cavg)
Multiple - dosed PK steps | After collecting blood samples from the last participant, up to 30 days
  -- Trough plasma concentration at steady state (Ctrough)
Multiple - dosed PK design | After collecting blood samples from the last participant, up to 30 days
  -- Time to reach peak concentration at steady state (Tmax,ss)
Multiple - dosed PK plan | After collecting blood samples from the last participant, up to 30 days
  -- Area under the concentration-time curve within time span t1 to t2 at steady state (AUCt1→t2,ss)
Multiple - dosed PK program | After collecting blood samples from the last participant, up to 30 days
  -- AUC in 1 dosing interval (AUCτ) at steady state
Multiple - dosed PK process | After collecting blood samples from the last participant, up to 30 days
  -- Terminal half-life at steady state (t1/2,ss)
Multiple - dosed PK arrangement | After collecting blood samples from the last participant, up to 30 days
  -- Apparent oral clearance at steady state (CL/Fss)
Multiple - dosed PK planning | After collecting blood samples from the last participant, up to 30 days
  -- Apparent volume of distribution after oral administration at steady state (Vd/Fss)
Assessment of effect duration for IBUMR | After collecting blood samples from the last participant, up to 30 days
  -- For the plasma ibuprofen concentration of IBUMR at steady state, the time to drop to the Ctrough of IBURed-600mg will be calculated.
Evaluation of duration of IBUMR effect | After collecting blood samples from the last participant, up to 30 days
  -- Percentage of the test drug-treated subjects with higher or equal plasma ibuprofen concentrations at 12-hour at steady state (C12,ss) compared to the Ctrough of IBURed-600mg will be calculated.
Incidence of treatment-emergent adverse events (safety and tolerability) | After collecting blood samples from the last participant, up to 60 days
  Incidence of AEs and SAEs
safety and tolerability | After collecting blood samples from the last participant, up to 60 days
  incidence of abnormal Physical examination
Incidence of treatment-emergent adverse events | After collecting blood samples from the last participant, up to 60 days
  abnormal Vital signs
Incidence of sudden adverse events (safety and tolerability) | After collecting blood samples from the last participant, up to 60 days
  abnormal laboratory tests results
Incidence of treatment-induced adverse events (safety and tolerability) | After collecting blood samples from the last participant, up to 60 days
  abnormal 12-lead ECG exams

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Che Liu, M.D, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taiwan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert KS, Gernaat CM. Pharmacokinetics of ibuprofen. Am J Med. 1984 Jul 13;77(1A):40-6. doi: 10.1016/s0002-9343(84)80017-0. PMID 6465162
- [Background] Albert KS, Gillespie WR, Wagner JG, Pau A, Lockwood GF. Effects of age on the clinical pharmacokinetics of ibuprofen. Am J Med. 1984 Jul 13;77(1A):47-50. doi: 10.1016/s0002-9343(84)80018-2. PMID 6380280
- [Background] Barkin RL, Buvanendran A. Focus on the COX-1 and COX-2 agents: renal events of nonsteroidal and anti-inflammatory drugs-NSAIDs. Am J Ther. 2004 Mar-Apr;11(2):124-9. doi: 10.1097/00045391-200403000-00007. PMID 14999364
- [Background] Davies NM. Clinical pharmacokinetics of ibuprofen. The first 30 years. Clin Pharmacokinet. 1998 Feb;34(2):101-54. doi: 10.2165/00003088-199834020-00002. PMID 9515184
- [Background] Goldberg DS, McGee SJ. Pain as a global public health priority. BMC Public Health. 2011 Oct 6;11:770. doi: 10.1186/1471-2458-11-770. PMID 21978149
- [Background] Legg T, Paluch E, Jayawardena S. Single- and Multiple-Dose Pharmacokinetics of Immediate-Release/Extended-Release Ibuprofen Tablets. Clin Pharmacol Drug Dev. 2017 Jan;6(1):36-43. doi: 10.1002/cpdd.288. Epub 2016 Sep 22. PMID 27364900
- [Background] Devarakonda K, Kostenbader K, Giuliani MJ, Young JL. Single- and multiple-dose pharmacokinetics of biphasic immediate-release/extended-release hydrocodone bitartrate/acetaminophen (MNK-155) compared with immediate-release hydrocodone bitartrate/ibuprofen and immediate-release tramadol HCl/acetaminophen. J Pain Res. 2015 Sep 30;8:647-56. doi: 10.2147/JPR.S83416. eCollection 2015. PMID 26508885
- [Background] O'Connor TP, Anderson AM, Lennox B, Muldoon C. A novel sustained-release formulation of ibuprofen provides effective once-daily therapy in the treatment of rheumatoid arthritis and osteoarthritis. Br J Clin Pract. 1993 Jan-Feb;47(1):10-3. PMID 8461240
- [Background] Varrassi G, Pergolizzi JV, Dowling P, Paladini A. Ibuprofen Safety at the Golden Anniversary: Are all NSAIDs the Same? A Narrative Review. Adv Ther. 2020 Jan;37(1):61-82. doi: 10.1007/s12325-019-01144-9. Epub 2019 Nov 8. PMID 31705437
- [Background] Volans G, Hartley V, McCrea S, Monaghan J. Non-opioid analgesic poisoning. Clin Med (Lond). 2003 Mar-Apr;3(2):119-23. doi: 10.7861/clinmedicine.3-2-119. No abstract available. PMID 12737366